CLINICAL TRIAL: NCT04038463
Title: Effects of Resistance Training in Body Composition and Body Image Perception of Women Throughout the Menstrual Cycle
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pandemic
Sponsor: Southern Illinois University Edwardsville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 160
Record Dates: First submitted 2019-05-21; First posted 2019-07-30 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2019-07

CONDITIONS: Body Image Disturbance
Keywords: Menstrual Cycle; Resistance Training; Body Composition; Intervention; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early Follicular Phase (EFP) (Experimental): The group will engage in the Resistance Training intervention on the fourth day of their menstrual cycle, which will correlate with the middle of the early follicular phase (EFP).
  Interventions: Behavioral: EFP
- Late Follicular Phase (LFP) (Experimental): The group will engage in the Resistance Training intervention on the eleventh day of their menstrual cycle, which will correlate with the middle of the late follicular phase (LFP).
  Interventions: Behavioral: LFP
- Early Luteal Phase (ELP) (Experimental): The group will engage in the Resistance Training intervention on the eighteenth of their menstrual cycle, which will correlate with the middle of the early luteal phase (ELP).
  Interventions: Behavioral: ELP
- Late Luteal Phase (LLP) (Experimental): The group will engage in the Resistance Training intervention on the twenty-fifth day of their menstrual cycle, which will correlate with the middle of the late luteal phase (LLP).
  Interventions: Behavioral: LLP

INTERVENTIONS:
Behavioral: EFP — This intervention will take place on day 4 of the participants' menstrual cycle. This will correspond to the mid-point of the early follicular phase (EFP).
  Arms: Early Follicular Phase (EFP)
Behavioral: LFP — The intervention will take place on day 8 of the participants' menstrual cycle. This will correspond to the mid-point of the late follicular phase (LFP).
  Arms: Late Follicular Phase (LFP)
Behavioral: ELP — The intervention will take place on day 18 of the participants' menstrual cycle. This will correspond to the mid-point of the early luteal phase (ELP).
  Arms: Early Luteal Phase (ELP)
Behavioral: LLP — The intervention will take place on day 25 of the participants' menstrual cycle. This will correspond to the mid-point of the late luteal phase (LLP).
  Arms: Late Luteal Phase (LLP)

SUMMARY:
The objective of this research study is two-fold, 1) to determine if body composition and body image perception are affected through the different phases of the menstrual cycle, and 2) if an acute session of resistance training can have different effects depending on the menstrual cycle phase.

DETAILED DESCRIPTION:
The purpose of the research is to establish whether body composition and body image perception are affected throughout the different phases of the menstrual cycle and if the perception can be modified through resistance training. To the best of our knowledge, only one study has analyzed the effects of the menstrual cycle on body image perception. However, research analyzing the effects of the menstrual cycle on both body image perception and, body composition is lacking. Furthermore, research in the effects of resistance training on menstrual cycle-related changes on both perceived and measured body composition are inexistent. Findings from this study have the potential to increase the knowledge about resistance training's effects in modulating body image perception throughout the menstrual cycle. Further understanding of these responses may set the groundwork to develop exercise intervention programs to reduce the risk of developing more serious mental conditions linked to unhealthy body image perception.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Sedentary or Active
* 18.5-34.9 kg/m2 BMI
* Normal menstrual cycle defined as 28 to 30 days and a duration of 3 to 7 days
* Age range is 18-45 years old
* The inclusion of other participants may alter the results as an increase in body fat has been linked to known changes in different hormonal levels and those changes might influence substrate utilization
* Changes in the hormonal status of pre-menopausal women may appear without symptoms
* Younger females also display variations in their hormones since they are going through the process of development

Exclusion Criteria:

* Previous physiological and mental health history
* Pregnant females
* Males
* Irregular menstrual cycle, menstrual dysfunction or unusual sex hormone levels
* Musculoskeletal injuries
* Contraceptives, a medication that alters hormonal or cardio-respiratory responses
* Pre-menopausal symptoms
* On moderate to high-intensity exercise regime more than 2 days/week

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be female and have normal menstrual cycles.
Enrollment: 6 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Body Image Perception through questionnaire | Through study completion: an average of 1 month
  Participants will be distributed the Multidimensional Body-Self Relations Questionnaire-Appearance Scale (MBSRQ-AS) to measure their body image perceptions.
Body Image Perception through drawing scale | Through study completion: an average of 1 month
  Participants will be distributed the Contour Drawing Rating Scale to measure their body image perception.
Barriers to Weight Control | Through study completion: an average of 1 month
  Participants will be distributed the Survey of Barriers to Weight Control to measure their body image perception.
Fat Mass in Kilograms | Through study completion: an average of 1 month
  We will measure fat mass using the Dual-Energy Xray Absorptiometry (DXA)
Lean Body Mass in Kilograms | Through study completion: an average of 1 month
  We will measure lean body mass using the Dual-Energy Xray Absorptiometry (DXA)
Relative Body Fat | Through study completion: an average of 1 month
  We will measure relative body fat (percentage) using the Dual-Energy Xray Absorptiometry (DXA)

SECONDARY OUTCOMES:
Bench Press One Repetition Maximum | At baseline: 1 assessment point prior randomization
  Participants muscular strength will be assessed by a one-repetition (1RM) on bench press
Leg Press One Repetition Maximum | At baseline: 1 assessment point prior randomization
  Participants lower body muscular strength will be assessed by a one-repetition (1RM) on leg press
Dietary habits | Before each exercise session: 1 assessment point on each menstrual cycle phase
  The participants diet will be recorded using the ASA-24h recall
Estrogen (Estradiol) levels | Before each exercise session: 1 assessment point on each menstrual cycle phase
  Blood will be drawn from the participants for assessment of the estrogen hormone
Progesterone levels | Before each exercise session: 1 assessment point on each menstrual cycle phase
  Blood will be drawn from the participants for assessment of the progesterone hormone

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernandez del Valle, PhD, Principal Investigator — Southern Illinois University Edwardsville
Locations (1):
- Southern Illinois University Edwardsville, Edwardsville, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided